CLINICAL TRIAL: NCT06637020
Title: A Randomized, Double-blind, Placebo-controlled, Phase Ib Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Subcutaneous (SC) Doses of HDM1005 Injection in Overweight or Obese Subjects
Brief Title: Phase Ib Clinical Study of HDM1005 Injection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou Zhongmei Huadong Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: HDM1005-102
Record Dates: First submitted 2024-05-31; First posted 2024-10-15 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2024-07

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- HDM1005 injection dose level 1 (Experimental): HDM1005 injection or pleacebo dose level 1 qw subcutaneous injection, 4weeks
  Interventions: Drug: HDM1005 injection or placebo
- HDM1005 injection dose level 2 (Experimental): HDM1005 injection or pleacebo dose level 2 qw subcutaneous injection, 4weeks
  Interventions: Drug: HDM1005 injection or placebo
- HDM1005 injection dose level 3 (Experimental): HDM1005 injection or pleacebo dose level 3 qw subcutaneous injection, 4weeks
  Interventions: Drug: HDM1005 injection or placebo
- HDM1005 injection dose level 4 (Experimental): HDM1005 injection or pleacebo dose level 3 qw subcutaneously administered once weekly, for 2 times; subsequently increased to dose level 4 once weekly for 2 times.
  Interventions: Drug: HDM1005 injection or placebo

INTERVENTIONS:
Drug: HDM1005 injection or placebo — Within each cohort, subjects are randomized in a 4:1 ratio to receive either HDM1005 injection or placebo subcutaneously.
  Other Names: HDM1005

SUMMARY:
This study is a randomized, double-blind, placebo-controlled, multiple-dose, dose-escalation study in overweight or obese subjects to evaluate the safety, tolerability, pharmacokinetic (PK), and pharmacodynamic (PD) characteristics of HDM1005 injection in overweight or obese subjects.

DETAILED DESCRIPTION:
This study is designed to consist of 5 dose cohorts, with 10 subjects in each cohort. Within each cohort, subjects are randomized in a 4:1 ratio to receive either HDM1005 injection or placebo subcutaneously. The proposed dose cohorts are as follows: cohort a (0.5 mg), cohort b (1.0 mg), cohort c (2.0 mg), cohort d (4.0 mg), cohort e (8.0 mg). Cohorts d,e will use a titration method to gradually reach the target dose. After obtaining safety and tolerability data for at least 14 days following multiple ascending dose (MAD) in the previous dose cohort, the dose to be administered and titration strategy for the next dose cohort are jointly determined by the investigator and the sponsor. Administration is allowed in the higher dose cohort only if the data from the lower dose cohort is indicative of safety. If necessary, the sponsor may continue to explore higher dose cohorts with the agreement of both the investigator and the sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18 to 65 years old (inclusive).
* BMI >27.0 kg/m² and < 40.0 kg/m² at screening and randomization.
* Blood pressure < 160/100 mmHg and pulse rate between 50-100 bpm (inclusive) at screening.
* Female subjects of childbearing potential must have used and agreed to continue using effective contraception methods for at least 14 days prior to signing the ICF and up to 2 months after dosing, and have no plans to have children or donate eggs. Male subjects must have no plans to have children or donate sperm from the date of signing the ICF to 4 months after dosing, and they must agree to use effective contraception methods.
* Able to understand the procedures and methods used in the study, voluntarily sign the ICF, and willing to strictly adhere to the requirements of the clinical trial protocol to complete the relevant procedures.

Exclusion criteria

Subjects who meet any of the following criteria will be excluded:

* Within 3 months before screening, subjects' body weight changed by ≥5%
* Previously diagnosed with type 1, type 2, or another type of diabetes
* Diagnosis of overweight or obesity due to other diseases or medications
* History or family history of medullary thyroid carcinoma, thyroid C-cell hyperplasia, or multiple endocrine adenomatosis type 2
* As determined by the investigator, the subjects have co-existing diseases or conditions that affect gastric emptying or gastrointestinal nutrient absorption.
* Cardiovascular and cerebrovascular diseases, gastrointestinal diseases, diabetes mellitus, medullary thyroid cancer, thyroid C cell hyperplasia, multiple endocrine adenomatosis type 2, chronic pancreatitis, and malignant tumors with obvious clinical significance were present; And any respiratory, neurological, urogenital, hematological, or endocrine disorders that may affect the safety of the subject or the findings of the study
* Any malignancy within 5 years prior to signing the ICF (except for basal cell carcinoma that has received curative treatment and is considered cured)
* Patients who have undergone major surgery within 3 months before signing the ICF, or who plan to undergo surgery during the study period
* Previous or combined depression or other mental disorders
* Known intolerance or allergy to any component of the investigational drug or GLP-1 receptor (GLP-1R) agonists; Or have a history of severe drug allergies
* Use of GLP-1R agonists within 6 months before signing the ICF
* Drugs that have been used within 3 months before signing ICF and have been determined by researchers to significantly affect weight and glucose
* For subjects taking lipid-lowering drugs, the dose of lipid-lowering drugs was not stable within 30 days before signing the ICF
* Participated in any clinical trial within 30 days prior to randomization or within 5 half-lives (whichever is older) after the last administration of the investigational drug in the clinical trial (except those who signed ICF and did not receive drug or device intervention)
* Any of the auxiliary test indicators during the screening period meets the following criteria:

  a) Hemoglobin <100g/L for women and < 110g/L for men; b) ALT>2.0x upper limit of normal (ULN), or AST>2.0x ULN, or ALP>1.5x ULN, or TBIL>1.5x ULN (Subjects with Gilbert's syndrome can participate in this study if DBIL≤ULN); c) HbA1c≥6.5%, or fasting blood glucose ≥7.0 mmol/L or ≤3.9 mmol/L; d) Triglyceride >5.6 mmol/L; e) calcitonin ≥20 ng/L; f) Thyroid stimulating hormone >6.0 mIU/L or <0.4 mIU/L g) blood amylase or lipase >ULN; h)eGFR < 90 mL/min/1.73m2; i) QTcF Male >450ms, female >470ms
* People tested positive for infectious diseases
* Habitual smokers, alcoholics and drug abusers
* Blood donors within 3 months prior to randomization
* Pregnant or lactating women
* The Investigator considers that the subject is not suitable to participate in any other circumstances of the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-06-20 (Actual); Primary Completion 2024-12-27 (Actual); Study Completion 2025-02-14 (Actual)

PRIMARY OUTCOMES:
The incidence, severity, and causality of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) | Signing informed until day 57
  Safety Outcomes . The incidence, severity, and causality of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) occurring during the study period; TEAEs leading to early study termination; TEAEs leading to death, etc.

SECONDARY OUTCOMES:
area under the concentration- time curve from time zero to time t (AUC0-t). | Before the first dose to 672 hours after the last dose
  PK parameter: area under the concentration- time curve from time zero to time t (AUC0-t).

OTHER OUTCOMES:
Changes of weight in kilogram | Baseline to day 29
BMI in kg/m^2 | Baseline to day 29
Changes of glucose | Baseline to day 29
Change of blood pressure | Baseline to day 29
Change of Total cholesterol (blood lipid ) | Baseline to day 29

CONTACTS AND LOCATIONS:
Overall Officials: Wei Hu, Doctor, Principal Investigator — The Second Hospital of Anhui Medical University
Locations (1):
- The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China